CLINICAL TRIAL: NCT05063058
Title: Feasibility Study of Biomarker-driven Therapy Based on a Comprehensive Molecular Analysis of Tumor Tissue and Blood Collections in Melanoma
Brief Title: Biomarker-driven Therapy for Melanoma
Acronym: TREAT20plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Max-Planck Institut (Unknown); Alacris (Unknown)
Responsible Party: Principal Investigator, Ulrich Keilholz, Director Charité Comprehensive Cancer Center, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TREAT20plus
Record Dates: First submitted 2021-08-26; First posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Molecular guided therapy (Experimental)
  Interventions: Drug: Molecular guided therapy

INTERVENTIONS:
Drug: Molecular guided therapy — Biomarker-driven therapy according to recommandations of the precision oncology tumor board including MEK Inhibitors (Trametinib 2 mg/d, Selumetinib 75 mg 2/d), MET Inhibitors (Crizotinib 250 mg 2/d, or Cabozantinib 60mg/d), RAS Inhibitor (Sorafenib 400 mg 2/d), Cell cycle Inhibitor (Palbociclib 125 mg/d) and Checkpoint Inhibitor (Nivolumab 240 mg every 2 weeks).

SUMMARY:
Patients included will undergo biopsy and the molecular analysis will be discussed at the institutional molecular tumor board. The recommandation of the molecular tumor board will be provided to the physician in charge of the patient for final treatment desicion.

The main endpoints are the number of patients with actionable molecular alterations, the number of patients with a treatment recommendation, the number of patients receiving the recommended therapy, overall survival of the patients treated according to recommendations or not. For patients treated according to the recommendations: Response rate and progression free survival at 6 months according to RECIST criteria.

DETAILED DESCRIPTION:
Eligible patients have to have a histologically proven metastatic melanoma failing standard treatments. Other inclusion criteria included age ≥ 18 years; Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2; life expectancy ≥ 24weeks; adequate renal, liver, and bone marrow functions. Previous therapy with intravenous chemotherapy, immunotherapy or major surgery at least 4 weeks before inclusion was allowed. Patients were excluded if they had a history of cardiac disease or metastatic brain or meningeal tumors. The study is approved by the institutional research ethics board.

Molecular analysis is performed at the Max Planck Institute for Molecular Genetics Berlin and a comprehensive report is made available with 4-8 weeks. The molecular tumor board interprets the data and transforms them into treatment recommendations by identifying and prioritizing predictive biomarkers. The recommendations rely on the definition of evidence levels attributed to every single aberration and the interdisciplinary discussion of the aberrations with regard to patient situation, availability of drugs, and clinical trials. The recommendations are transmitted to the physician in charge of the patient for the final decision to treat or not the patient accordingly.

The main endpoints are the number of patients with actionable molecular alterations, the number of patients with a treatment recommendation, the number of patients receiving the recommended therapy, overall survival of patients treated according to recommendations or not.

For patients treated according to the recommendations: Response rate and progression free survival at 6 months according to RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven metastatic melanoma failing standard treatments
* age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* life expectancy ≥ 24 weeks
* adequate renal, liver, and bone marrow functions

Exclusion Criteria:

- history of cardiac disease or metastatic brain or meningeal tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Feasibility (actionable molecular alterations) | Through study completion over 5 years
  number of patients with actionable molecular alterations
Feasibility (number of patients with a treatment recommendation) | Through study completion over 5 years
  number of patients with a treatment recommendation
Feasibility (number of patients receiving the recommended therapy) | Through study completion over 5 years
  number of patients receiving the recommended therapy

SECONDARY OUTCOMES:
Overall survival | 5 years
  Overall survival
Response rate | 1 year
  Response rate of the patients treated according to the recommendations
Progression free survival at 6 months according to RECIST criteria | up to 6 months
  PFS according to RECIST criteria for the patients treated according to the recommendations